CLINICAL TRIAL: NCT04958772
Title: Clinical Trials Phase I, Single-Centric, Open, Randomized, Crossed, For Comparative Evaluation Of The Pharmacokinetic And Pharmacodynamic Profile Of The Filgrastim Injectable Solution, In Relation To The Comparison Granulokine®, Ltda. After Subcutaneous Multiple Administration In Healthy Participants
Brief Title: Biosimilarity Study of Subcutaneous Filgrastim in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Megalabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LATIM
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Filgrastim Megalabs (Experimental): Filgrastim Megalabs injectable 5 μg/Kg/day in a single subcutaneous application during 5 days
  Interventions: Biological: Filgrastim Megalabs; Biological: Granulokine
- Granulokine (Active Comparator): Granulokine injectable 5 μg/Kg/day in a single subcutaneous application during 5 days
  Interventions: Biological: Filgrastim Megalabs; Biological: Granulokine

INTERVENTIONS:
Biological: Filgrastim Megalabs — Filgrastim Megalabs 5 μg/Kg/day, subcutaneous single dose
Biological: Granulokine — Granulokine 5 μg/Kg/day, subcutaneous single dose

SUMMARY:
This study will compare the pharmacokinetics and pharmacodynamics, after single subcutaneous application, in healthy men, between filgrastim formulation, produced by Megalabs (test product) and Granulokine® (reference product) Amgen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy eligible participants able to read, understand and sign the latest version of the Informed Consent Form (ICF) approved by the Research Ethics Committee (CEP)
* Males aged between 18 and 55 years
* Be characterized as a healthy research participant, based on medical history general physical examination and vital signs, laboratory tests and electrocardiogram (ECG),
* Not indicating any evidence of disease
* Body weight between 60-100 kg
* Body Mass Index (BMI) ≥ 18.5 and ≤ 29.9 Kg / m2
* Negative test for coronavirus

Exclusion Criteria:

* Present one or more flu-like symptoms such as: fever (body temperature greater than or equal to 37.8 ° C), cough, dyspnoea, myalgia and fatigue, respiratory symptoms, gastrointestinal symptoms (such as diarrhea) within 7 days prior to the hospitalization period (all periods)
* Direct and significant medical contact with people who tested positive for coronavirus testing within 14 days prior to the hospitalization period (all periods)
* Living in the same household as people who are in the risk group with the worst prognosis for coronavirus infection, such as individuals over 60, individuals with respiratory problems, immunosuppressed or those with chronic diseases, such as heart or diabetes (all periods)
* Participants diagnosed with malignant disease in the last 5 years, with the exception of successfully treated basal cell carcinoma
* Participants with a previous diagnosis of severe asthma, sickle cell anemia, idiopathic urticaria or anaphylaxis
* Participants with chronic diseases and, therefore, who regularly use medications
* Being a smoker or quitting less than 6 months ago
* Participants who consume more than 5 cups of tea or coffee a day and who cannot - abstain during the trial period
* History of alcohol and illicit drug abuse
* Electrocardiogram (ECG) findings that, at the investigator's discretion, may compromise participation in the trial
* History or presence of gastrointestinal or liver diseases or any other condition that interferes with the absorption, distribution, excretion or metabolism of the drug
* Use of lithium 2 weeks before and / or after medication administration
* Participants who are hypersensitive or contraindicated to use any of the components of the formulation
* Research participants who have participated in clinical trial protocols in the last 12 (twelve) months (Resolution CNS 251, of August 7, 1997, item III, subitem J)
* Have donated blood (> 500 mL) or have undergone major surgery in the 3 (three) months preceding the date of signing the informed consent form
* Have received any vaccine in the 3 (three) months preceding the date of signing the informed consent form

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of AUC 0-t in healthy volunteers for test and reference. | 17 days
Evaluation of Cmax in healthy volunteers for test and reference. | 17 days
Evaluation of absolute neutrophil count (ANC) in healthy volunteers for test and reference. | 17 days

SECONDARY OUTCOMES:
Evaluation of CD34+ count for test and reference | 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Satish Kumar, MD, Principal Investigator — Azidus Principal Investigator

IPD SHARING:
Plan to Share IPD: No